CLINICAL TRIAL: NCT00004802
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Dichlorphenamide for Periodic Paralyses and Associated Sodium Channel Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Ohio State University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11958; OSU-92H0173
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: Paralysis, Hyperkalemic Periodic; Hypokalemic Periodic Paralysis; Paramyotonia Congenita
Keywords: neurologic and psychiatric disorders; periodic paralysis; rare disease
MeSH Terms: conditions — Paralysis, Hyperkalemic Periodic; Hypokalemic Periodic Paralysis; Myotonic Disorders; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Dichlorphenamide

INTERVENTIONS:
Drug: dichlorphenamide

SUMMARY:
OBJECTIVES:

I. Assess the efficacy of dichlorphenamide in the treatment of episodic weakness attacks in patients with hyperkalemic periodic paralysis, paramyotonia congenita with periodic paralysis, and hypokalemic periodic paralysis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution and diagnosis.

The weekly attack rate is determined during an 8-week assessment prior to therapy initiation and at crossover.

Patients are randomly assigned to oral dichlorphenamide (DCP) or placebo for 9 weeks and then cross to the alternate treatment. Patients on DCP at baseline continue on the same dose; those on acetazolamide (ACZ) at baseline receive a DCP dose equivalent to one fifth of the ACZ dose.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Hypokalemic periodic paralysis Typical clinical profile Normal serum thyroxine Hypokalemia during spontaneous or glucose-induced paralytic attack in subject or affected family member

Periodic paralysis associated with sodium channel 17q alpha-subunit, e.g.:

* Hyperkalemic periodic paralysis with or without myotonia
* Paramyotonia congenita with periodic paralysis

Distinct, regular episodes of weakness at least once a week and no more than 3 times a day

No history of worsening symptoms with carbonic anhydrase inhibitor

No history of life-threatening weakness episodes prior to treatment

No atypical periodic paralysis without demonstrable 17q alpha-subunit defect

--Prior/Concurrent Therapy--

No requirement for the following agents, unless for periodic paralysis:

* Diuretics
* Antiepileptics
* Antiarrhythmics
* Magnesium supplements
* Steroids
* Calcium supplements
* Beta-blockers
* Potassium supplements
* Calcium channel blockers

--Patient Characteristics--

Hepatic: No hepatic disease

Renal:

* No renal failure
* No nephrolithiasis

Cardiovascular:

* No heart disease
* No cardiac arrhythmia

Pulmonary: No restrictive or obstructive lung disease

Other:

* No active thyroid disease
* No pregnant women

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64
Dates: Start 1992-06

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, Study Chair — Ohio State University